CLINICAL TRIAL: NCT05019209
Title: Chamber Exposure with House Dust Mite (HDM) or Allergen-free Air in Atopic Drmatitis Patients with HDM Sensitization to Investigate the Role of Aeroallergen Exposure on Skin Responses and T Cell Immunology
Brief Title: Skin Responses and T Cell Immunology After House Dust Mite Exposure in Sensitized Atopic Dermatitis Patients
Acronym: CODES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, MD, Prof. Dr. Jens M Hohlfeld, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-06 CODES
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis; House Dust Mite Allergy
MeSH Terms: conditions — Dermatitis, Atopic; Dust Mite Allergy | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Intervention Model Description: All subjects are exposed to house dust mite and allergen-free air in the same sequence. Subjects are blinded to the sequence of house dust mite and allergen-free air exposures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exposure to saline-dissolved house dust mite allergen and allergen-free air (Experimental): Subjects are blinded to the sequence of interventions in the allergen challenge chamber (ACC). Overall, subjects will be in the ACC 4 times during the study. Of those, exposure to allergen-free air and HDM is allocated in a 2:2 ratio.
  Interventions: Drug: House Dust Mite Allergen; Other: Allergen-free air

INTERVENTIONS:
Drug: House Dust Mite Allergen — D. pteronyssinus lyophilisate dissolved in 5% sodium chloride solution, spray dried
Other: Allergen-free air — No allergen added to room ventilation of allergen challenge chamber

SUMMARY:
The present study investigates the reaction of the skin upon exposure to house dust mite (HDM) in patients with atopic dermatitis who have antibodies against HDM in the blood. A further aim is to assess nasal symptoms after exposure to HDM in an allergen challenge chamber and compare the results with data from previous studies.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic skin disease characterized by a relapsing course and typical clinical manifestation with itchy, eczematous lesions. The majority of AD patients reveals elevated IgE serum levels (> 100kU / L), which classifies the disease as extrinsic AD. Mostly, the IgE is directed against aeroallergens like pollen and house dust mite (HDM). These allergens may contribute pronouncedly to the relapsing character of the disease.

Of note, it was already shown in the 1920s that avoiding aeroallergens by sleeping in an allergen-free chamber has a positive influence not only on the symptoms of asthma but also on the skin condition in AD patients. However, a recent study was the first showing that challenge chamber exposure to airborne grass pollen allergens can cause a clinical worsening of the skin condition in sensitized AD patients. These standardized settings in the Fraunhofer Allergen Challenge Chamber can conduce as a model for the investigation of the impact on other allergens on AD patients.

For the perennial allergen HDM, Sager et al. investigated the epicutaneous application of HDM allergens in sensitized AD patients. It led to an aggravation of the eczematous lesions through a T-cell-mediated reaction. The binding of the HDM allergen to specific IgE-Fc receptors on Langerhans cells leads to the proliferation of specific T cells in the skin and a proinflammatory signaling. Until now, however, airborne HDM allergen exposure has not been shown to cause aggravation of AD in any controlled setting. This study aims to answer the question of the extent to which standardized exposure of AD patients with HDM has an impact on objective, subjective and in vitro disease parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Male and female subjects, aged 18-65 years. Women will be considered for inclusion if they are:
3. Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing.
4. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
5. Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the start of the study until at least 72 hours after the last study visit -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
6. Positive IgE level for HDM of at least CAP FEIA class 3 (≥3,50 kU/l) at screening or in previous year.
7. Atopic dermatitis fulfilling the UK criteria of AD
8. SCORAD index between 20 and 50 points.
9. Positive self-history regarding poor skin condition during fall and winter months and allergic rhinitis and/or conjunctivitis in situations of significant HDM exposure (e.g., dusting).
10. FEV1 ≥ 80% pred. at screening.
11. Total Nasal Symptom Score (TNSS) of ≤ 3 prior to entering the chamber at visit 2.
12. Smokers or non-smokers.
13. BMI ≥18 and ≤ 35.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, vital signs or lung function at screening visit , which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease.
3. Asthma other than mild asthma which is treated with short acting beta-2-agonists only and which is controlled according to the current GINA guidelines
4. Subject with concomitant allergies to seasonal aeroallergens which become active (i.e., grass, trees, weeds, rye; defined as being symptomatic to aeroallergens within the past 2 years or within the past 2 allergy seasons) during the individual study participation.
5. Positive HIV-1/2Ab, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCV-Ab) test at screening or test not performed.
6. Treatment with medication that might interfere with rescue medication for anaphylactic reactions (e.g. beta blocker).
7. Topical steroid treatment (wash out phase: 2 weeks before day 1)
8. Topical calcineurin inhibitor treatment (wash out phase 2 weeks before day 1)
9. UV radiation treatment (wash out phase 4 weeks before day 1)
10. Systemic immunosuppression treatment (steroids, biologics, e.g. dupilumab, JAK-Inhibitors, cyclosporine, azathioprine, Mycophenolat Mofetil (MMF); wash out phase 4 weeks and 3 months, respectively, before day 1.
11. Treatment with antihistamines (wash out phase 1 week).
12. Unstable AD during Screening (SCORAD difference of >10 points from Visit 1 to Visit 2)
13. Diastolic blood pressure above 95 mmHg.
14. Acute respiratory infection 2 weeks prior to screening visit.
15. Alcohol or drug abuse within 12 month prior to screening.
16. Regular daily consumption of more than 1 liter of usual beer or the equivalent quantity of approximately 40 g of alcohol in another form.
17. Participation in another clinical trial 30 days prior to enrollment.
18. There is a risk of non-compliance with study procedures.
19. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
20. History of an acute infection four weeks prior to the informed consent visit.
21. Subject has received previous immunotherapy treatment with any HDM allergen within 3 years prior to screening.
22. Subject is receiving ongoing treatment with any specific immunotherapy for other allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Change in the objective SCORAD | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  SCORAD is an established score taking severity of typical lesions, the extent of involvement of the skin and the subjective items itch and sleeplessness into account. The subjective symptoms will be assessed referring to the period of time of the past three days.
  The objective SCORAD is based on the calculation of the SCORAD mentioned above, but without the subjective parameters itch and sleeplessness

SECONDARY OUTCOMES:
Difference of change in local SCORAD | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  SCORAD is an established score taking severity of typical lesions, the extent of involvement of the skin and the subjective items itch and sleeplessness into account. The subjective symptoms will be assessed referring to the period of time of the past three days.
  The objective SCORAD is based on the calculation of the SCORAD mentioned above, but without the subjective parameters itch and sleeplessness
Change in SCORAD index | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  SCORAD is an established score taking severity of typical lesions, the extent of involvement of the skin and the subjective items itch and sleeplessness into account. The subjective symptoms will be assessed referring to the period of time of the past three days.
  The objective SCORAD is based on the calculation of the SCORAD mentioned above, but without the subjective parameters itch and sleeplessness
Change of itch (VAS) | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  The subjects rate their actual skin itch on a visual analog scale (VAS). The VAS is an unmarked line with a length of 10cm. The left end of the line is labeled "no itch" and the right end is labeled "worst itch imaginable". Each time the subjects assess their itch they have to mark the line at the position they feel their symptoms are at this moment in relation to the symptoms described at both ends of the line
Increase of the rescue medication use | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  Rescue medications are class II topical glucocoticosteroids and topical calcineurin inhibitors
Change of the DLQI | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  The dermatological life quality index (DLQI) is a valid measuring instrument that represents the health-related quality of life in skin diseases. Each of the questions is rated with 0-3 points, from which the total value is added
Change of IGA | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  The Investigator's Global Assessment scale (IGA) score provides information about the overall appearance of the lesions at a specific point in time. It is not necessary that all characteristics are included under Morphological Description. The score is divided into 5 levels from clear to severe.
Change of EASI | Baseline assessment on Day 4 and immediately after exposure in allergen challenge chamber
  The Eczema Area and Severity Index (EASI) is another score evaluating the Skin in AD patients. The body surface is divided according to percentage. To assess the severity of the lesions, they are analyzed in detail in terms of erythema, infiltration, excoriation and lichenification. Values between 0 and 72 can be calculated.
Differences of skin related severity scores between clean- and HDM exposure | Day 1 to Day 6
  skin behaviour rating between study groups
Difference of AUC2-4hTNSS between clean- and HDM exposure | Day 1 to Day 6
  Mean over two hours of subjective nasal symptoms between study groups
Difference of AUC2-4hTNSS between HDM exposure | Day 1 to Day 6
  Mean over two hours of subjective nasal symptoms between exposure sessions
Difference of maximum TNSS between clean-air and HDM exposure | Day 1 to Day 6
  Maximum degree of subjective nasal symptoms between study groups
Difference of maximum TNSS between HDM exposure | Day 1 to Day 6
  Nasal symptoms will be evaluated by the subject prior to and every 20 minutes during allergen challenge according to the 4 point severity scale including nasal congestion, rhinorrhea, nasal itching and sneezing. Each symptom can be scored from 0 (no symptoms) to 3 (severe symptoms). Scores range from 0 to 12.
Difference of nasal secretion weight per hour between clean-air and HDM exposure | Day 1 to Day 6
  Subjects will receive pre-weighed sachets of handkerchiefs which will be weighed again after exposure in the allergen challenge chamber.
Difference of nasal secretion weight per hour between HDM exposure | Day 1 to Day 6
  Subjects will receive pre-weighed sachets of handkerchiefs which will be weighed again after exposure in the allergen challenge chamber.
Change in nasal secretion weight between pre-challenge and the sum of post challenge nasal secretion weights of both allergen-free air exposures | Day 1 to Day 6
  Subjects will receive pre-weighed sachets of handkerchiefs which will be weighed again after exposure in the allergen challenge chamber.

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer ITEM
Locations (2):
- Germany (2):
  - Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Lower Saxony
  - Hannover Medical School, Department of Dermatology and Allergy, Hanover, Lower Saxony

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werfel T, Allam JP, Biedermann T, Eyerich K, Gilles S, Guttman-Yassky E, Hoetzenecker W, Knol E, Simon HU, Wollenberg A, Bieber T, Lauener R, Schmid-Grendelmeier P, Traidl-Hoffmann C, Akdis CA. Cellular and molecular immunologic mechanisms in patients with atopic dermatitis. J Allergy Clin Immunol. 2016 Aug;138(2):336-49. doi: 10.1016/j.jaci.2016.06.010. PMID 27497276
- [Background] Werfel T, Heratizadeh A, Niebuhr M, Kapp A, Roesner LM, Karch A, Erpenbeck VJ, Losche C, Jung T, Krug N, Badorrek P, Hohlfeld JM. Exacerbation of atopic dermatitis on grass pollen exposure in an environmental challenge chamber. J Allergy Clin Immunol. 2015 Jul;136(1):96-103.e9. doi: 10.1016/j.jaci.2015.04.015. Epub 2015 Jun 1. PMID 26044854
- [Background] Sager N, Feldmann A, Schilling G, Kreitsch P, Neumann C. House dust mite-specific T cells in the skin of subjects with atopic dermatitis: frequency and lymphokine profile in the allergen patch test. J Allergy Clin Immunol. 1992 Apr;89(4):801-10. doi: 10.1016/0091-6749(92)90434-4. PMID 1373161